CLINICAL TRIAL: NCT00477750
Title: Phase I/II Trial of Melphalan, Prednisone Plus Lenalidomide in Patients With Newly Diagnosed Multiple Myeloma Who Are Not Candidates for Stem Cell Transplant
Brief Title: Melphalan, Prednisone, and Lenalidomide in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546642; P30CA015083 (NIH); MC038A (Other: Mayo Clinic Cancer Center); 2387-04 (Other: Mayo Clinic IRB); RV-MM-PI-025 (Other: Celgene protocol)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2015-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Melphalan; Prednisone

ARMS (1):
- Treatment (Lenalidomide, Melphalan, Prednisone) (Experimental): Intervention: Drug: lenalidomide Dose determined by Phase I treatment schedule. Taken orally days 1-21 every 28 days until progression
  Intervention: Drug: melphalan Dose determined by Phase I treatment schedule. Taken orally days 1-4 every 28 days until progression
  Intervention: Drug: prednisone 60mg/m^2, orally days 1-4 every 28 days until progression
  Interventions: Drug: lenalidomide; Drug: melphalan; Drug: prednisone

INTERVENTIONS:
Drug: lenalidomide — Phase I - dose escalating: 5mg level -1, 10mg level 0, 10mg level 1, 15mg level 2, 20mg level 3, 25mg level 4, orally days 1-21 every 28 days until progression
  Phase II - 10 mg orally days 1-21 every 28 days until progression
Drug: melphalan — Phase I - dose escalating: 5mg/m^2 dose level -1, 5 mg/m^2 dose level 0, 8 mg/m^2 dose level 1 - 4, daily x 4 orally days every 28 days until progression
  Phase II - 5mg/m^2 orally days 1-4 every 28 days until progression
Drug: prednisone — 60mg/m^2, orally days 1-4 every 28 days until progression

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, prednisone, and lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of melphalan and lenalidomide when given together with prednisone and to see how well they work in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of melphalan and lenalidomide in combination with prednisone in patients with newly diagnosed multiple myeloma.
* Determine the response rate in patients treated with this regimen. Secondary
* Determine the toxicity of this regimen in these patients. OUTLINE: This is a dose-escalation study of melphalan and lenalidomide followed by a phase II study.
* Phase I: Patients receive oral melphalan and oral prednisone daily on days 1-4. Patients also receive oral lenalidomide daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of melphalan and lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oral melphalan and oral lenalidomide as in phase I at the MTD. Patients also receive oral prednisone as in phase I. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Newly diagnosed disease
  * Requires treatment, in the judgment of the treating physician
  * Not a candidate for (or patient declines) autologous stem cell transplantation
* Meets 1 of the following criteria:

  * Measurable disease, defined by any of the following:

    * Serum monoclonal protein ≥ 1 g/dL
    * Urine protein monoclonal light chain ≥ 200 mg/24 hours by electrophoresis
    * Measurable serum free light chains ≥ 10 mg/dL, kappa or lambda, AND κ/λ ratio is abnormal (if serum and urine are not measurable as defined above)
  * Evaluable disease, defined as monoclonal bone marrow plasmacytosis ≥ 30%

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 3.0 mg/dL
* Platelet count ≥ 100,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception, including ≥ 1 highly effective method, ≥ 4 weeks before and during study treatment
* No uncontrolled infection
* No peripheral neuropathy ≥ grade 2
* No serious medical condition, laboratory abnormality, or psychiatric illness that would preclude study compliance
* No other active malignancy except for nonmelanoma skin cancer or carcinoma in situ

  - Prior malignancy allowed if treated with curative intent and is free of disease for a period appropriate for that cancer
* No known hypersensitivity to thalidomide
* No known HIV positivity
* No infectious hepatitis A, B or C
* No history of deep vein thrombosis or other medical condition requiring the use of warfarin
* Able to take daily prophylactic acetylsalicylic acid (81 or 325 mg)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy for treatment of multiple myeloma
* No prior lenalidomide
* No other concurrent anticancer agents or treatments
* No concurrent steroids except prednisone ≤ 20 mg/day (or the equivalent) for concurrent illness or adrenal replacement therapy
* No other concurrent investigational therapy or agent for treatment of multiple myeloma
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2013-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Roy, MD, FACP, Study Chair — Mayo Clinic; Philip R. Greipp, MD, Principal Investigator — Mayo Clinic; Craig B. Reeder, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was as Phase I/II trial. There were 7 patients recruited to the Phase I portion; no patients qualified for the Phase II portion. Twenty-six (26) patients were recruited for the Phase II portion. Results presented here are on the 26 Phase II patients.
Groups:
- Treatment (Lenalidomide, Melphalan, Prednisone): Intervention: Drug: lenalidomide 10 mg orally days 1-21 every 28 days until progression
  Intervention: Drug: melphalan 5mg/m^2 orally days 1-4 every 28 days until progression
  Intervention: Drug: prednisone 60mg/m^2, orally days 1-4 every 28 days until progression
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Started | 26
Completed | 15
Not Completed | 11
Not completed — Currently Receiving Treatment | 11

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 73.5 [64 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 26
Durie-Salmon Stage at Diagnosis [Number; unit: participants]
  I - Low Cell Mass | 1
  II - Intermediate Cell Mass | 11
  III - High Cell Mass | 11
  unknown | 3
Parameter of Hematologic Response - Serum M-spike >= 1g/dL [Number; unit: participants]
  Yes | 20
  No | 6
Parameter of Hematologic Response - Serum Immunoglobulin Free Light Chain >= 10mg/dL [Number; unit: participants]
  Yes | 12
  No | 14
Parameter of Hematologic Response - Urine M-spike >= 200 mg/24 hours [Number; unit: participants]
  Yes | 6
  No | 20
Parameter of Hematologic Response - None (non-secretory myeloma, bone marrow only) [Number; unit: participants]
  Yes | 0
  No | 26

OUTCOME MEASURES:

1. Primary Outcome: Patients With Overall Confirmed Response
Description: Response that was confirmed on 2 consecutive evaluations.>
  * Complete Response (CR): Complete disappearance of M-protein from serum and urine on immunofixations, normalization of Free Light Chain (FLC) ratio and <=5% plasma cells in bone marrow>
  * Very Good Partial Response (VGPR): >=90% reduction in serum M-spike, Urine M-spike <100mg per 24 hours>
  * Partial Response (PR): >=50% reduction in serum M-spike, Urine M-spike >=90% reduction or < 200mg per 24 hours, or >=50% decrease in difference between involved and uninvolved FLC levels or 50% decrease in bone marrow plasma cells
Time Frame: Every cycle during treatment
Measure: Number; unit: participants
Groups:
- Treatment (Lenalidomide, Melphalan, Prednisone): Intervention: Drug: lenalidomide 10 mg orally days 1-21 every 28 days until progression> > Intervention: Drug: melphalan 5mg/m^2 orally days 1-4 every 28 days until progression>
  > Intervention: Drug: prednisone 60mg/m^2, orally days 1-4 every 28 days until progression
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 26
participants
  CR | 3
  VGPR | 5
  PR | 10

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression was defined as any one or more of the following:
  An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
Time Frame: registration to progressive disease (up to 3 years)
Population: Phase 2 patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 26
months | 21.4 [15.3 to 23.5]

3. Secondary Outcome: Overall Survival (OS) at 3 Years
Description: OS was defined as the time from registration to death due to any cause. Patients who were alive were censored at date of last follow-up. The overall survival at 3 years (a percentage) is reported below.
Time Frame: registration to death (up to 3 years)
Population: Phase 2 patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 26
percentage of patients | 58 [42 to 80]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was calculated from documentation of first response to date of progression in the subset of patients who responded. Patients without progression were censored at the date of last tumor evaluation.
Time Frame: from first response to progression or death (up to 3 years)
Population: Phase 2 Patients who had a response of PR or better are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 18
months | 16.3 [14.3 to 26.4]

5. Secondary Outcome: Percentage of Participants With Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (v3)
Description: The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Every cycle during treatment up to 3 years
Population: Patients who experienced an adverse event that is at least possibly related are included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Number analyzed (Participants) | 3
percentage of patients
  Grade 3 | 33
  Grade 4 | 67
  Grade 5 | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Lenalidomide, Melphalan, Prednisone)
Serious Adverse Events (participants affected / at risk) | 7/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Melphalan, Prednisone) (N=26)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Melphalan, Prednisone) (N=26)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 (103)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (12)
Edema limbs (General disorders) | 11 (27)
Fatigue (General disorders) | 21 (63)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 2 (5)
Hypersensitivity (Immune system disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (5)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 6 (13)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 18 (58)
Platelet count decreased (Investigations) | 18 (70)
Blood glucose increased (Metabolism and nutrition disorders) | 15 (32)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (8)
Syncope (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (14)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes